CLINICAL TRIAL: NCT02947230
Title: Evaluating the Impact of the McMaster Optimal Aging Portal on Knowledge, Behavioural Intentions and Health Behaviours Related to Physical Mobility
Brief Title: Evaluating the Impact of the McMaster Optimal Aging Portal on Physical Mobility Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-04
Record Dates: First submitted 2016-10-21; First posted 2016-10-27 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2019-03

CONDITIONS: Mobility Limitation
Keywords: Mobility; Aging; Knowledge Translation; Physical Activity
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored Knowledge Translation (Experimental): During the 12-week KT intervention, intervention group participants will have access to the Portal and will receive mobility-focused weekly email alerts including blog posts and evidence summaries relevant to mobility and be invited to follow a Twitter and Facebook feed; a unique hashtag will be created to identify and collate relevant mobility information.
  Interventions: Other: Tailored Knowledge Translation
- Control group (No Intervention): Participants in the control group will have access to the Portal in a 'self-serve' fashion. These participants will be able to browse the Portal, subscribe to email alerts, follow social media, etc. but will not receive the tailored mobility intervention.

INTERVENTIONS:
Other: Tailored Knowledge Translation — Tailored knowledge translation strategies specific to maintaining and increasing physical mobility with age.
  Arms: Tailored Knowledge Translation

SUMMARY:
The McMaster Optimal Aging Portal (the Portal) was launched in 2014 to increase public access to trustworthy health information. The Portal helps readers to access evidence-based resources; identify trustworthy messages; and understand scientific findings. Now the investigators want to know whether using the Portal changes what people know and do to stay healthy and mobile.

This project will help us to:

1. Understand how middle aged and older adults (age 40+) use the Portal to obtain information about maintaining and improving mobility
2. Evaluate whether use of the Portal results in a change in knowledge about maintaining and improving mobility, or change in lifestyle behaviours that may help maintain or improve mobility with age.

DETAILED DESCRIPTION:
Physically active lifestyles are important for health aging, but most Canadians do not meet published physical activity guidelines. This may be in part due to lack of access to evidence-based information on mobility and aging, and knowledge of strategies to maintain or improve mobility with age. The McMaster Optimal Aging Portal (the Portal) was launched in 2014 to increase public access to trustworthy health information. Now the investigators want to know if easy-to-understand evidence-based messages change what people know and do to stay healthy and mobile.

Sequential, explanatory mixed-methods design consisting of a two-armed randomized controlled trial and a qualitative process study to explore quantitative findings in depth.

Consent forms and a baseline survey will be sent to all interested participants. Following baseline data collection, participants will be stratified by previous Portal use, and randomized to the Knowledge Translation (KT) intervention or control group. During the 12-week KT intervention, intervention group participants will have access to the Portal and will receive mobility- focused weekly email alerts including blog posts and evidence summaries relevant to mobility and be invited to follow a Twitter and Facebook feed; a unique hashtag will be created to identify and collate relevant mobility information. Control group participants will be able to access the Portal in a 'self-serve' fashion, but will not receive targeted KT strategies.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking

Exclusion Criteria:

* None

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Website analytics | 12 weeks
  Understanding participant engagement with the Portal and knowledge translation strategies
Email analytics | 12 weeks
  Understanding participant engagement with the Portal and knowledge translation strategies
Google analytics | 12 weeks
  Understanding participant engagement with the Portal and knowledge translation strategies

SECONDARY OUTCOMES:
Knowledge Questionnaire | 12 weeks, 3 months post-intervention
  Participants knowledge of mobility recommendations and guidelines
Beliefs Questionnaire | 12 weeks, 3 months post-intervention
  Participants beliefs about the importance of maintaining and improving mobility for health
Intentions Questionnaire | 12 weeks, 3 months post-intervention
  Participants intentions to engage in lifestyle behaviours related to maintaining or improving mobility
Rapid Assessment of Physical Activity | 12 weeks, 3 months post-intervention
  To quantify self-reported physical activity
Manty Preclinical Mobility Disability Scale | 12 weeks, 3 months post-intervention
  Mobility limitation

OTHER OUTCOMES:
Participant satisfaction | 12 weeks
  Collected using qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Dobbins, RN, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neil-Sztramko S, Smith-Turchyn J, Richardson J, Dobbins M. Impact of a Knowledge Translation Intervention on Physical Activity and Mobility in Older Adults (the Move4Age Study): Randomized Controlled Trial. J Med Internet Res. 2020 Feb 11;22(2):e15125. doi: 10.2196/15125. PMID 32044750
- [Result] Neil-Sztramko SE, Smith-Turchyn J, Richardson J, Dobbins M. A Mobility-Focused Knowledge Translation Randomized Controlled Trial to Improve Physical Activity: Process Evaluation of the Move4Age Study. J Med Internet Res. 2019 Jun 20;21(6):e13965. doi: 10.2196/13965. PMID 31223121